CLINICAL TRIAL: NCT04478461
Title: A Phase Ia Clinical Trial to Assess Safety, Tolerability, and Pharmacokinetics of a Recombinant Humanized Anti-PD-1 Monoclonal Antibody (MW11) for Injection in Patients With Advanced Solid Tumors
Brief Title: Safety, Tolerability, and Pharmacokinetics of MW11 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MW11-2019-CP101
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MW11 injection (Experimental): 1, 3, 10 mg/kg and maybe an additional fixed dose (e.g., to evaluate 200 mg or other fixed dose as RP2D). The drug is scheduled to be administrated Q3W.
  Interventions: Drug: PD-1 monoclonal antibody

INTERVENTIONS:
Drug: PD-1 monoclonal antibody — The enrollment mainly depends on "3+3" principle. A total of 3 or 4 dose groups will be evaluated during the dose escalation period: 1, 3, 10 mg/kg, and maybe an additional fixed dose (e.g., to evaluate 200 mg or other fixed dose as RP2D). The drug is scheduled to be administrated Q3W
  Other Names: MW11 injection

SUMMARY:
This is a phase Ia, single-center, open label, dose escalation clinical study to evaluate the safety, tolerability, pharmacokinetics, immunogenicity and anti-tumor efficacy of MW11 (a recombinant humanized anti-PD-1 monoclonal antibody) for injection in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The enrollment mainly depends on "3+3" principle. A total of 3 or 4 dose groups will be evaluated during the dose escalation period: 1, 3, 10 mg/kg, and maybe an additional fixed dose (e.g., to evaluate 200 mg or other fixed dose as RP2D). The drug is scheduled to be administrated Q3W. Actual dose increments or dosing frequency may be adjusted according to PK data and safety of MW11. Safety, tolerability, and DLT will be assessed within 3 weeks (21 days) after initial administration. Anti-tumor efficacy will be assessed every 6 weeks during the first 24 weeks and every 12 weeks ever since. The study will be divided into screening period and treatment period. The drug administration will be continued until the investigators consider that the subjects will no longer benefit from the treatment, or the subjects meet intolerable toxicity, or the subjects withdraw the informed consent, or disease progression occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged from 18 to 75 (including 18 and 75).
2. Pathological diagnosis of advanced or metastatic solid tumors.
3. Advanced solid tumors that are progressed after standard antitumor therapy and can not accept or refuse to receive standard treatment.
4. The ECOG score is 0 or 1.
5. The subjects are expected to survive at least 3 months.
6. Subjects must have at least 1 measurable lesion according to response evaluation criteria in solid tumors RECIST V1.1. The measurable lesion must be absent from the previous radiotherapy area or have progressed radiologically 4 weeks after radiotherapy.
7. The subjects have proper organ and hematopoietic function, no serious heart, lung, liver, renal function abnormalities or immune deficiency according to the following laboratory tests:

   Hematology: Absolute neutrophils count (ANC) ≥ 1.5×109/L, platelet ≥ 100×109/L, hemoglobin ≥ 90g/L.

   Renal function: serum creatinine ≤ 1.5 times the upper limit of normal value (ULN) or creatinine clearance ≥ 50 mL/ min (Chockcroft-Gault formula was used for creatinine clearance).

   Liver function: AST and ALT ≤ 2.5 times ULN(AST and ALT ≤ 5 times ULN in patients with liver cancer or liver metastasis; serum total bilirubin (TBIL) ≤ 1.5 times ULN; alkaline phosphatase ≤ 1.5 times ULN(alkaline phosphatase≤ 5 times ULN in patients with liver cancer or liver metastasis, or patients with bone metastasis).

   Coagulation function: international normalized ratio (INR) ≤ 2 times ULN, or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN (except for the subjects who are receiving anticoagulant therapy).
8. Male subjects with fertility and female subjects of reproductive age are willing to take effective contraceptive measures from the signing of informed consent until 6 months after the last dose of drug administration. Female subjects of reproductive age (before menopause and women after menopause within 2 years) must have negative blood pregnancy test results within 7 days before the first drug administration.
9. Subjects sign informed consent voluntarily, to make sure they understand the study and are willing to follow and able to complete all trial procedures.

Exclusion Criteria:

Prior or current medical conditions:

1. Previous history of other malignant tumors (any malignant tumor other than the tumor species treated in this study), except that the tumor has been cured for ≥ 2 years before screening and treatment is not required during the study period.
2. Brain metastases.
3. Prior adverse reactions failed to recover to CTCAE V5.0 grade score ≤ 1, with the exception of residual hair loss effect.
4. Fluid accumulations in the body cavity (pleural effusion, ascites, pericardial effusion, etc.) that are not well controlled and require local treatment or repeated drainage.
5. With active, or history of autoimmune diseases that may recur (E.G. systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.) , or high-risk patients, such as those who have received an organ transplant and require immunosuppressive therapy. But subjects with the following diseases are allowed to be enrolled:

   Subjects with type I diabetes whose condition is stable after receiving fixed dose of insulin (HgbA1C ≤ 6.5%).

   Autoimmune hypothyroidism requiring only hormone replacement therapy. Vitiligo, or skin diseases that do not require systemic treatment (such as eczema that accounts for less than 10% of the body surface, psoriasis without ophthalmic symptoms, etc.).
6. Sudden onset of pulmonary disease, Interstitial lung disease or pneumonia, or other uncontrolled systemic disease including diabetes, pulmonary fibrosis, acute lung disease, cardiovascular disease including hypertension (for example, LVEF ≤50% or NYHA ≥ III) , with the exception of locally interstitial pneumonia due to radiotherapy.
7. Subjects infected by human immunodeficiency virus (HIV), or with other acquired or congenital immunodeficiency diseases, or with a history of organ transplantation or stem cell transplantation.
8. Subjects with active tuberculosis infection within 5 years before enrollment.
9. Subjects who were seriously infected within 4 weeks prior to the first drug administration, or who had any signs or symptoms of active infection within 2 weeks priorly, or who required antibiotic treatment within 2 weeks priorly (except for the prophylactic antibiotics); or patients who had unexplained fever >38.5℃ before the first drug administration (subject with fever caused by tumor can be enrolled according to the investigator's judgment).

   Prior medication or treatment:
10. Patients who have received anti-PD-1 or PD-L1 antibody therapy or have received any other antibody/drug (such as CTLA-4) therapy targeting T-cell co-regulatory proteins (immune checkpoint) within 12 weeks prior to the first drug administration of the study.
11. Subjects who have received anti-tumor therapy except:

    The interval between systemic radiotherapy and the first drug administration of this study is ≥ 4 weeks, and the interval of local or bone metastasis radiotherapy is ≥ 2 weeks. No radiological agents were taken within 8 weeks prior to the first drug administration of this study.

    Prior chemotherapy interval ≥ 4 weeks, immunotherapy, biological therapy (tumor vaccine, cytokines, or growth factors that control cancer), or approved targeted and other therapies, must be completed before the first drug administration in this study, and the interval must be no less than 5 half-lives or at least 6 weeks (whichever is longer).

    TCM treatment should be completed at least 14 days before the first drug administration in this study.
12. Subjects require systemic corticosteroids (the dosage is equivalent to >10 mg prednisone per day) or other immunosuppressive drugs within 14 days prior to enrollment. Enrollment is allowed in the following cases:

    Subjects are allowed to use topical or inhaled glucocorticoids. Subjects are allowed to use glucocorticoids in short-term (≤ 7 days) for the prevention or treatment of non-autoimmune allergic diseases that do not occur frequently.
13. Subjects who have received immunotherapy and had an immune-related adverse event (irAE) level ≥ 3.

    History of allergies, general conditions and others:
14. A subject is known to have had a prior severe allergic reaction to a macromolecular protein preparation/monoclonal antibody or any component of the tested drug (CTCAE V5.0 rating is greater than level 3).
15. Subjects with chronic hepatitis B/ active hepatitis C/ syphilis. However, hepatitis B virus carriers, stable hepatitis B after drug treatment (DNA ≤ normal value), and cured hepatitis C patients (HCV RNA negative) can be enrolled.
16. Subjects who participated in other drug clinical trials within 4 weeks prior to enrollment.
17. Subjects who had major surgery within 4 weeks prior to screening or who are expected to have major surgery during the study period (including the 28-day screening period).
18. Subjects with history of alcohol, drug or substance abuse in the last 1 year.
19. Subjects with clear history of neurological or psychiatric disorders, such as epilepsy, dementia, or poor compliance.
20. Females who are pregnant or breastfeeding.
21. Subjects with any other medical condition that is considered to affect the subject's safety.
22. The subjects that the investigator considers unsuitable for the study due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2023-01-05 (Estimated); Study Completion 2023-02-02 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE ) | 2 years
  safety evaluation
Severity Adverse Event (SAE) | 2 years
  safety evaluation

SECONDARY OUTCOMES:
Elimination half life（t1/2） | 2 years
  safety/efficacy evaluation
Area under the concentration-time curve（AUC） | 2 years
  safety/efficacy evaluation
volume of distribution （Vz） | 2 years
  safety/efficacy evaluation
Plasma Clearance （CL） | 2 years
  safety/efficacy evaluation
Maximum Plasma Concentration（Cmax） | 2 years
  safety/efficacy evaluation
Time to maximum plasma concentration（Tmax） | 2 years
  safety/efficacy evaluation
Objective remission rate (ORR) | 2 years
  efficacy evaluation
Disease control rate (DCR) | 2 years
  efficacy evaluation
Duration of remission (DOR) | 2 years
  efficacy evaluation
Progression free survival (PFS) | 2 years
  efficacy evaluation
Overall survival (OS) | 2 years
  efficacy evaluation
Number of Participants with positive anti drug antibody (ADA) | 2 years
  safety evaluation
Number of Participants with positive neutralizing antibody (Nab) | 2 years
  safety evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, professor, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China